CLINICAL TRIAL: NCT05609357
Title: The Feasibility and Safety of Head-up Cardiopulmonary Resuscitation in Patients With Non-traumatic Cardiac Arrest: Single Center Research
Brief Title: The Feasibility and Safety of Head-up Cardiopulmonary Resuscitation in Patients With Non-traumatic Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202204040DIND
Record Dates: First submitted 2022-10-19; First posted 2022-11-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; Head-up Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head-up Cardiopulmonary Resuscitation (Experimental)
  Interventions: Device: Head-up Cardiopulmonary Resuscitation

INTERVENTIONS:
Device: Head-up Cardiopulmonary Resuscitation — Elevate patient's head to 30 degrees by EleGARD System during cardiopulmonary resuscitation

SUMMARY:
Head up CPR with impedance threshold device(ITD) and active compression-decompression (ACD) has been proved to improve both cerebral and coronary perfusion pressure during resuscitation in animal models. Increased rates of Spontaneous Circulation (ROSC) were also observed in cardiac arrest patients.

The goal of this clinical trial is to learn about the feasibility and safety of Head-up Cardiopulmonary Resuscitation in patients with non-traumatic cardiac arrest. Participants will be received head-up CPR during resuscitation. The main question it aims to answer is if there is any adverse or unfavorable event during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic cardiac arrest
* Age ≥ 20

Exclusion Criteria:

* Trauma
* Age < 20
* Pregnancy
* Irreversible death (e.g. liver mortis, rigor mortis, decapitation, transection and decomposition)
* Disorder of cervical spine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and portion of participants with serious or non-serious adverse event | Up to 1 day
  e.g. event of fall, failure of intubation

SECONDARY OUTCOMES:
Number and portion of participants with repeated CPR | up to 1 day
Number and portion of participants with survival to emergency department discharge | up to 1 day
Number and portion of participants with sustained return of spontaneous circulation | Up to 1 day
  sustained ROSC ≥ 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ting Chen, Principal Investigator — National Taiwan University Hospital; Chien-Hua Huang, Principal Investigator — National Taiwan University Hospital; Min-Shan Tsai, Principal Investigator — National Taiwan University Hospital; Chih-Hsien Lin, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No